CLINICAL TRIAL: NCT02387255
Title: Magnetic Resonance Elastography in Patients With Abdominal Aortic Aneurysms
Acronym: AAA-MRE
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Arunark Kolipaka, Associate Professor, Ohio State University
Other Study IDs: 2013H0416
Record Dates: First submitted 2015-02-19; First posted 2015-03-12 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect a small aortic tissue sample for biomechanical testing from patients undergoing standard of care surgical repair of their abdominal aortic aneurysm.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Volunteers: 60 normal volunteers will be recruited. Each volunteer will undergo a single MRE scan (with Resoundant driver System ) of their abdominal aorta.
  Interventions: Device: Resoundant Driver System
- Patients with AAA: Fifty to sixty five patients with AAA will be recruited. These patients will undergo MRE (with Resoundant driver system) of their AAA every six months for three years, or until the study ends or until the time of surgical repair or death due to rupture of AAA or other causes.
  Interventions: Device: Resoundant Driver System
- Open Surgical Repair Patients: Fifty to sixty five patients patients undergoing open surgical repair will be recruited and undergo MRE (with Resoundant driver system) prior to surgery
  Interventions: Device: Resoundant Driver System

INTERVENTIONS:
Device: Resoundant Driver System — This device is used to generate vibrations at the area of interest. The device has an active driver, a loud speaker sitting outside the scanner area, and a passive driver, which is shaped like a silicone paddle, which is secured with velcro straps to the area being imaged. Sound waves from the active driver travel through a tube attached to the passive driver and generate vibrations, images of which are captured by the MR scanner.
  Other Names: Driver

SUMMARY:
The main objective of this study is to utilize Magnetic Resonance Elastography (MRE) to determine tissue stiffness of abdominal aortic aneurysms (AAA). For patients with AAA, MRE is a more sensitive and superior method of determining the risk for rupture of AAA based on stiffness estimates when compared to the current, crude method of assessing risk based on measurement of the diameter of the aneurysm. The investigators will also validate the stiffness estimates against gold standard i.e. mechanical testing and histopathology only AAA patients undergoing AAA surgery.

DETAILED DESCRIPTION:
Currently, MRE is a clinical tool used to assess hepatic fibrosis at many institutions. MRE is superior to invasive techniques (i.e. biopsies) and mechanical testing in that it is noninvasive and can be performed in vivo under physiologic conditions. MRE could make diagnosing stiffness widely available and could revolutionize the diagnosis and treatment of numerous other diseases affecting stiffness of soft tissues.

Aortic wall "stiffness" is a fundamental biomechanical parameter that reflects the structural integrity of normal and aneurysmal aortic tissue. AAAs enlarge over time leading to sudden rupture and death in up to 90% of patients. Surgical or endovascular aneurysm repair (EVAR) is recommended for AAAs > 5.5 cm in diameter. However, previous studies have reported a high percentage (13%) of smaller AAAs (<5 cm) go on to rupture, and an even higher percentage (60%) of larger AAAs (>5 cm) remain stable. Despite the poor prognostic value of aortic diameter, it is still the primary parameter used to time surgical repair. It is known that changes in stiffness of AAA can reveal important information on extra-cellular matrix content; a key factor in the pathophysiological development of AAA and the risk for rupture. A non-invasive, spatially resolved estimate of aortic stiffness may provide a superior determinant of the risk for rupture compared to the currently used anatomical measures. The relationship between non-invasively measured wall stiffness (WS) and the structural integrity of the aortic wall must be further elucidated. Therefore, aortic MRE can be used as a noninvasive tool to estimate the stiffness of AAAs and can provide superior diagnostic and prognostic information in patients with developing AAA disease.

Entry to this study is open to men and women aged 18 years and older, and to all racial and ethnic subgroups. Two separate groups of patients with AAA will be recruited. One group will be patients who have been diagnosed with AAA and are monitored to observe the size of the AAA. The other group is comprised of patients who are scheduled for surgical repair of AAA.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to lie flat on their back in the scanner for up to 60 minutes
* Must be able to hold breath for up to 15 seconds

Exclusion Criteria:

* Patients who are claustrophobic
* Patients who are pregnant
* Patients with any unapproved, non-MRI save metal/devices in or on their body

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal volunteers are control group
  2. Patients who are being monitored for diameter of AAA
  3. Patients who will undergo surgical repair of AAA
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2014-10; Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
MRE-Derived Shear Stiffness in kPa | Upto 36 months at every 6 months
  Use of MRE stiffness estimates to determine rupture

CONTACTS AND LOCATIONS:
Overall Officials: Arunark Kolipaka, PhD, Principal Investigator — The Ohio State University Medical Center Dept. of Radiology
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States